CLINICAL TRIAL: NCT00577447
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Docosahexaenoic Acid Supplementation in Children With Autism
Brief Title: Docosahexaenoic Acid in the Treatment of Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Robert G. Voigt, MD/ Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 398-05
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Autism
Keywords: autism; omega-3 fatty acids; docosahexaenoic acid
MeSH Terms: conditions — Autistic Disorder | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): DHA supplemented group
  Interventions: Dietary Supplement: docosahexaenoic acid (DHA)
- 2 (Placebo Comparator): Placebo group
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: docosahexaenoic acid (DHA) — Capsule containing 200mg of DHA
  Arms: 1
Dietary Supplement: Placebo — Placebo capsule containing corn and soybean oil
  Arms: 2

SUMMARY:
The purpose of this study is to test the hypothesis that dietary supplementation with the omega-3 fatty acid docosahexaenoic acid (DHA) improves the behavior of children with autism.

DETAILED DESCRIPTION:
Autism is a neurodevelopmental disability with an increasing prevalence. Traditional medicine does not offer any cures for autism; thus, many parents of children with autism are attracted to complementary and alternative therapies, one of which is dietary supplementation with the long chain polyunsaturated omega-3 fatty acid, docosahexaenoic acid (DHA). DHA is a critical structural lipid of brain cell membranes and differences in brain DHA content may influence synaptic function, particularly in nutritionally-sensitive areas of the brain, such as the cerebellum and hippocampus, which may be brain structures involved in the etiology of autism. This study is a randomized, double-blind, placebo-controlled trial investigating whether DHA supplementation is an effective treatment for children with autism. Eighty children with autism will be randomized to receive 200mg of DHA or placebo for 6 months. Outcome variables will include total plasma fatty acid patterns and scores on parent and investigator-completed behavioral and developmental rating scales at baseline and after 3 and 6 months of supplementation. Differences between groups after 6 months will be evaluated using regression methods. Regression analysis will be used to detect correlations between plasma total fatty acid DHA contents and scores on the various outcome measures. Results from this study will either provide evidence for a breakthrough biomedical treatment alternative for children with autism or evidenced-based advice to desperate parents in regard to their choices of potential treatments for their children with autism

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for autistic disorder
* Age 3 to 10 years

Exclusion Criteria:

* Use of a dietary supplement containing DHA within 90 days of study inclusion
* Medical history of a disorder of lipid metabolism

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2005-10; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions-Improvement Scale | 6 months

SECONDARY OUTCOMES:
Child Development Inventory | 6 months
Behavior Assessment Scale for Children | 6 months
Aberrant Behavior Checklist | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Voigt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States